CLINICAL TRIAL: NCT00523731
Title: A Study of Blood-Borne Autologous Angiogenic Cells Precursors Therapy in Patients With Critical Limb Ischemia
Brief Title: ACPs in Severe PAD/CLI by Direct Intramuscular Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TheraVitae Ltd. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TV-003; ACPs-CLI
Record Dates: First submitted 2007-08-30; First posted 2007-08-31 (Estimated); Last update posted 2007-08-31 (Estimated); Status verified 2007-02

CONDITIONS: Peripheral Arterial Disease; Critical Limb Ischemia
Keywords: Stem cells; Rest pain; claudication; chronic ischemic or non-healing ulcers; Angiogenesis; no-option cases
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia; Intermittent Claudication | interventions — holo-(acyl-carrier-protein) synthase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Angiogenic Cell Precursors (ACPs) or Vescell TM

SUMMARY:
Study title: A Study of Blood-Borne Autologous Angiogenic Cell Precursors Therapy in Patients with Critical Limb Ischemia ( ACPs-CLI )

Principle Investigator: Assoc.Prof. Pramook Mutirangura,M.D. Head of Division of Vascular Surgery , Department of Surgery, Faculty of Medicine Siriraj Hospital , Mahidol University, BKK,Thailand

Study objective : To determine the safety and efficacy of intramuscular injection of blood-borne autologous ACPs in relieving symptoms of critical limb ischemia of patients treated with maximal medical therapy and don't have intravascular or operative revascularization option.

Study Design : A pilot study , a single center, a non-randomized, open-label trial.

Total expected no. of patients : 6 main selection criteria : A. Subjects will have one or more clinical indications diagnostic of CLI such as: distal extremity pain at rest that requires the subject to use analgesics for >2 weeks; or peripheral ischemic ulcer(s); or areas of gangrene ; or non-healing ischemic ulcers AND

B. Subjects will have one or more of the following hemodynamic indicators of severe peripheral arterial occlusive disease:

I. Ankle brachial index < 0.45 II. Toe brachial index < 0.35 III. TcPO2 / TcO2 of < 40 mmHg. C. The subject is a poor candidate for standard revascularization treatment for peripheral arterial disease, based on inadequate bypass conduit, or unfavorable anatomy D. Age 18 to 80 years

Investigational Product : At D-8 250 ml of blood drawn from the patients for production of autologous EPCs or ACPs (VescellTM). On D0 ,at least 1.5 million ACPs with viability >75 % suspended in 30 ml sterile cell culture medium will be injected 1.5 cm deep and 1.5 apart by a 23 -gauge needle into the gastrocnemius muscle of the leg chosen (ischemic leg) for treatment. For injection planning a grid of 10X10 cm will be prepared and in each point 1 ml of ACPs suspension will be injected.

The study consists of 4 periods: Screening ( D-14 to-9& D-8,Treatment(D0),Acute Safety follow-up (D1&D2),Chronic follow-up (D30 & D90)period ,total follow-up of each case is 3 months.

Evaluation criteria :

Safety : no.& duration of adverse event & serious adverse event Efficacy :Attenuate CLI patients symptoms (Rest pain,Pain-free walking distance,Ulcer size &Gangrene dimension and intensity)

DETAILED DESCRIPTION:
Six patients with Critical Limb Ischemia (CLI) or severe Peripheral Arterial Disease(PAD) will be enrolled, screened, treated with an injection of Blood-Borne Autologous Angiogenic Cell Precursors(ACPs) in to gastrocnemius of the ischemic leg by intramuscular under regional anesthesia. Following injection.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will have one or more clinical indications diagnostic of CLI such as: distal extremity pain at rest that requires the subject to use analgesics for >2 weeks; or peripheral ischemic ulcer(s); or areas of gangrene ; or non-healing ischemic ulcers AND
* Subjects will have one or more of the following hemodynamic indicators of severe peripheral arterial occlusive disease:

  * Ankle brachial index < 0.45
  * Toe brachial index < 0.35
  * TcPO2 / TcO2 of < 40 mmHg.
* The subject is a poor candidate for standard revascularization treatment options for peripheral arterial disease, based on inadequate bypass conduit, or unfavorable anatomy
* Age 18 to 80 years
* Male or non-pregnant, non-lactating female
* Informed consent obtained and consent form signed

Exclusion Criteria:

* Patient having on angiography a meaningful supra popliteal occlusion that may relate to symptoms of CLI.
* Subjects, who in the opinion of the investigator, have a vascular disease prognosis that indicates they would require a major amputation (at or above the ankle) within 4 weeks of start of treatment
* Patient who received blood transfusions during the previous 4 weeks (to exclude the potential of non-autologous ACPs in the harvested blood).
* Inability to communicate (that may interfere with the clinical evaluation of the patient)
* Major operation during the preceding 3 months
* Myocardial infarction or brain infarction or uncontrolled myocardial ischemia or persistent severe heart failure (EF< 25 %) during the preceding 3 months
* Significant valvular disease or after valve replacement during the preceding 3 months
* After heart transplantation
* Severe cardiomyopathy (EF < 25 %)
* Renal failure (creatinine > 2 mg/dl )
* Hepatic failure
* Anemia (lower than 11mg/dl.hemoglobin for female and lower than 12 mg/dl for male)
* Abnormal coagulation tests [platelets, PT (INR), PTT]
* Stroke within the preceding 3 years
* Malignancy within the preceding 3 years
* Concurrent chronic or acute infectious disease
* Severe concurrent medical disease (e.g., septicemia, HIV-1,2/HBV/HCV infections, poorly controlled insulin-dependent diabetes mellitus ; HBA1c >8 % and proliferative retinopathy , systemic lupus erythematosus, multiple sclerosis, amyotrophic lateral sclerosis)
* Chronic immunomodulating or cytotoxic drugs treatment
* Patients who have rectal temp. above 38.40C for 2 consecutive days
* Patient unlikely to be available for follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-01; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Safety | 3 months
Evaluate the safety of ACPs intramuscular injection | 3 months
Efficacy | 3 months
Attenuate CLI patients symptoms as | 3 months
Rest pain | 3 months
Pain-free walking distance | 3 months
Ulcer size | 3 months
Gangrene dimension and intensity | 3 months
Obtain evidence for improvement of tissue perfusion due to ACPs injection | 3 months

SECONDARY OUTCOMES:
Reduction of CLI patients hospitalization time. | 3 months
Decrease CLI patient amputation rate. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Pramook Mutirangura, M.D., Principal Investigator — Vascular Surgery Unit,Department of Surgery,Faculty of Medicine Siriraj Hospital,Mahidol University,BKK,Thailand
Locations (1):
- Dr. Valentin Fulga, Tel Viv, P.O.B.4049,Ness Ziona, Israel

REFERENCES:
- [Derived] Mutirangura P, Ruangsetakit C, Wongwanit C, Chinsakchai K, Porat Y, Belleli A, Czeiger D. Enhancing limb salvage by non-mobilized peripheral blood angiogenic cell precursors therapy in patients with critical limb ischemia. J Med Assoc Thai. 2009 Mar;92(3):320-7. PMID 19301723